CLINICAL TRIAL: NCT04940130
Title: Phase 2 Trial of Safety, Immunogenicity, and Efficacy Against Plasmodium Falciparum Malaria of PfSPZ Vaccine in Children in Mali
Brief Title: PfSPZ Vaccine Trial in Malian Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanaria Inc. (Industry)
Collaborators: Malaria Research and Training Center, Bamako, Mali (Other); University of the Sciences, Techniques and Technologies of Bamako (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MLSPZV5
Record Dates: First submitted 2021-06-03; First posted 2021-06-25 (Actual); Results first posted 2024-02-07 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2023-12

CONDITIONS: Malaria; Malaria,Falciparum
Keywords: PfSPZ Vaccine; Malaria; Plasmodium falciparum
MeSH Terms: conditions — Malaria; Malaria, Falciparum | interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: randomized, placebo controlled, with concurrent arms
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double-blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 (PfSPZ Vaccine) (Experimental): 134 children ages 6 - 10 will receive three doses of PfSPZ Vaccine (9.0x10^5 PfSPZ) via DVI at 1, 8, and 29 days
  Interventions: Biological: Sanaria® PfSPZ Vaccine
- Arm 2 (normal saline) (Placebo Comparator): 134 children ages 6 - 10 will receive normal saline via DVI at 1, 8, and 29 days
  Interventions: Other: Normal Saline

INTERVENTIONS:
Biological: Sanaria® PfSPZ Vaccine — non-adjuvanted, live (metabolically active), radiation-attenuated, non-replicating, whole sporozoite (SPZ) vaccine designed to prevent malaria infection caused by Plasmodium falciparum (Pf).
  Arms: Arm 1 (PfSPZ Vaccine)
Other: Normal Saline — placebo control- saline
  Arms: Arm 2 (normal saline)

SUMMARY:
In this randomized, double-blind, placebo-controlled trial, 268 healthy Malian children aged 6-10 years, residing in Bancoumana and surrounding villages, will be administered three doses of 9.0x10^5 Pf sporozoites (PfSPZ) of PfSPZ Vaccine (or placebo) at 1, 8, and 29-days using direct venous inoculation (DVI).

The study is composed of a single cohort with two arms (categorized by placebo control/experimental groups) designed to assess the safety, immunogenicity and protective efficacy of PfSPZ Vaccine.

All subjects will receive artemether-lumefantrine (AL) approximately 1- 2 weeks before the first dose of PfSPZ Vaccine or normal saline for clearance of Pf parasitemia. Vaccinated participants and non-immunized controls will be followed for safety and monitored for development of parasitemia through the natural malaria transmission season to estimate vaccine efficacy (VE).

DETAILED DESCRIPTION:
This phase 2 study will enroll healthy Malian children between 6 and 10 years of age residing in Bancoumana and surrounding villages to participate in a randomized, double blind, placebo- controlled study to assess the safety, immunogenicity and protective efficacy of PfSPZ Vaccine.

Participants will be immunized with a 3-dose series of 9.0 x10^5 PfSPZ of PfSPZ Vaccine or normal saline (placebo) at 1, 8, and 29 days. Subjects will be screened for eligibility for enrollment. Enrollment will begin with AL dosing approximately 1-2 weeks prior to their first dose of vaccine. Volunteers will be randomized into two arms (1 vaccine arm, 1 control arm) in a 1:1 ratio.

Vaccinated subjects and controls will then be followed for safety and assessment for malaria infection during the subsequent malaria transmission season.

268 children between the ages of 6 and 10 years old inclusive will be enrolled as follows:

Arm 1(PfSPZ Vaccine): (n = 134) children ages 6 - 10 will receive three doses of PfSPZ Vaccine (9.0x10^5 PfSPZ) via direct venous inoculation (DVI) at 1, 8, and 29 days

Arm 2 (normal saline): (n = 134) children ages 6 - 10 will receive normal saline via DVI at 1, 8, and 29 days All subjects will receive artemether-lumefantrine (AL) approximately 1- 2 weeks before the first dose of PfSPZ Vaccine or normal saline for clearance of Pf parasitemia.

Vaccinated participants and non-vaccinated controls will be monitored for development of Pf malaria with symptoms and Pf malaria (parasitemia) through the natural malaria transmission season to estimate vaccine efficacy (VE). During the surveillance period, both active and passive surveillance will be used to identify Pf malaria with symptoms. Blood smears will be made at any time a participant presents with a clinical syndrome consistent with malaria and read in real time, with all infections treated.

In addition, blood smears will be made every four weeks in all participants as active surveillance for Pf malaria (parasitemia). However, to avoid confounding the primary clinical endpoint, these blood smears will be read retrospectively at the end of the primary surveillance period.

Primary Case Definition:

Pf malaria with symptoms is defined as a positive thick blood smear at a density of >1000 parasites/uL (P/uL) plus:

* Measured auxiliary temperature ≥ 37.5 degrees Celsius or history of fever (subjective or objective) in the last 24 hours, or,
* Symptoms of malaria -

  * Verbal individual (individual able and willing to answer questions): A verbal individual is considered symptomatic if reporting at the time of evaluation at least two of the following symptoms/symptom groups: headache, chills and/or rigors, malaise and/or fatigue, dizziness and/or light-headedness, myalgias and/or arthralgias; or
  * Non-verbal individual (small child or any individual unable or unwilling to answer questions): A non-verbal individual is considered symptomatic if manifesting at the time of evaluation at least two of the following signs/sign groups: drowsiness, irritability and/or fussiness, inability and/or refusal to eat or drink, prostration; or
  * Any individual: Signs of severe malaria (e.g. impairment of consciousness, severe anemia, hemoglobinuria, acute kidney injury, etc.)

Secondary Case Definition:

Pf malaria with symptoms is defined as a positive thick blood smear at a density of > 0 P/uL plus:

* Measured axillary temperature ≥ 37.5 degrees Celsius or history of fever (subjective or objective) in the last 24 hours, or,
* Symptoms of malaria as defined in the primary case definition; or
* Meeting criteria for severe malaria

Pf malaria is defined as:

- At least one unambiguous asexual parasite on thick blood smear identified by two independent microscopists after each examining 0.50 μL of blood in a study participant

ELIGIBILITY:
Inclusion Criteria:

1. Parent(s) or guardian(s) willing and able to provide consent prior to initiation of any study procedures
2. Stated willingness of parent(s) or guardian(s) to comply with all study procedures and availability for the duration of the study
3. Malaria comprehension exam completed by parent(s) or guardian(s) and passed with a score of ≥80% or per investigator's discretion
4. Healthy children 6-10 years of age at enrollment (inclusive)
5. Parent(s) or guardian(s) are able to provide proof of identity to the satisfaction of the study clinician completing the enrollment process
6. Willing to have blood samples stored for future research

Exclusion Criteria:

1. Medical, behavioral, cognitive, or psychiatric disease that in the opinion of the investigator affects the ability of the participant's parent and/or legal guardian to understand and comply with the study protocol
2. Menstruating females (in order to avoid cultural implications of further assessing pregnancy potential i.e. sexual activity in this age group)
3. Hemoglobin (Hgb), WBC, absolute neutrophils, and platelets outside the local laboratory-defined limits of normal and ≥ Grade 2 (subjects may be included at the investigator's discretion for 'not clinically significant' abnormal values)
4. Alanine transaminase (ALT) or creatinine (Cr) level above the local laboratory-defined upper limit of normal and ≥ Grade 2 (subjects may be included at the investigator's discretion for 'not clinically significant' abnormal values)
5. Infected with human immunodeficiency virus (HIV), hepatitis B, or hepatitis C
6. Sickle cell disease by history
7. Taking or planning to take seasonal malaria chemoprophylaxis
8. Clinically significant abnormal electrocardiogram (ECG) such as abnormal QTc
9. History of receipt of the following:

   * Investigational malaria vaccine in the last 2 years
   * Immunoglobulins and/or blood products within 6 months of enrollment
   * Investigational product within 3 months of enrollment
   * Chronic (≥14 days) oral or IV corticosteroids (excluding topical or nasal) at immunosuppressive doses (i.e., prednisone ≥20 mg/day or equivalent) or immunosuppressive drugs within 30 days of enrollment
   * Live vaccine within 30 days of enrollment
   * Killed vaccine within 14 days of enrollment or planned receipt of a killed vaccine within 14 days of scheduled vaccination
10. Known medical problems:

    * Pre-existing autoimmune or antibody-mediated diseases (e.g. systemic lupus erythematosus, rheumatoid arthritis, multiple sclerosis, Sjögren's syndrome, or autoimmune thrombocytopenia)
    * Severe asthma (defined as asthma that is unstable or required emergent care, urgent care, hospitalization, or intubation during the past two years, or that has required the use of oral or parenteral corticosteroids at any time during the past two years)
    * Immunodeficiency disorder
    * Asplenia or functional asplenia
    * Diabetes
    * Deep venous thrombosis or thromboembolic event
    * Seizures (exception is simple febrile seizures during childhood)
11. Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, endocrine, rheumatologic, autoimmune, hematological, oncologic, or renal disease by history, physical examination, and/or laboratory studies

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 290 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-12-10 (Actual); Study Completion 2022-12-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Duffy, MD, Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID); Issaka Sagara, MD MSPH PhD, Principal Investigator — Malaria Research and Training Center
Locations (1):
- Malaria Research and Training Center, Bamako, Mali

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1 (PfSPZ Vaccine): Children ages 6 - 10 will receive three doses of PfSPZ Vaccine (9.0x10^5 PfSPZ) via direct venous inoculation (DVI) at 1, 8, and 29 days
  Sanaria® PfSPZ Vaccine: non-adjuvanted, live (metabolically active), radiation-attenuated, non-replicating, whole sporozoite (SPZ) vaccine designed to prevent malaria infection caused by Plasmodium falciparum (Pf).
- Arm 2 (Normal Saline): Children ages 6 - 10 will receive normal saline via DVI at 1, 8, and 29 days
  Normal Saline: placebo control- saline
- Enrolled With no Arm Assignment: Children ages 6 -10 were enrolled upon administration of AL treatment, but not assigned to a treatment arm (did not receive PfSPZ Vaccine nor Normal saline)
Period: Overall Study
Arm/Group | Arm 1 (PfSPZ Vaccine) | Arm 2 (Normal Saline) | Enrolled With no Arm Assignment
Started | 139 | 138 | 13
Completed | 138 | 137 | 0
Not Completed | 1 | 1 | 13
Not completed — Travel | 1 | 0 | 2
Not completed — Parent/Guardian withdrew consent | 0 | 1 | 7
Not completed — Adverse Event | 0 | 0 | 2
Not completed — Disease progression/treatment failure | 0 | 0 | 1
Not completed — Participant refusal | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 (PfSPZ Vaccine) | Arm 2 (Normal Saline) | Enrolled With no Arm Assignment | Total
Number analyzed (Participants) | 139 | 138 | 13 | 290
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 139 | 138 | 13 | 290
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 53 | 9 | 116
  Male | 85 | 85 | 4 | 174
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 139 | 138 | 13 | 290
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Mali | 139 | 138 | 13 | 290

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Possibly, Probably, or Definitely Related Serious Adverse Events (SAEs)
Description: Proportion of vaccinees compared to controls experiencing related SAEs from V1 to 26 weeks after V3
Time Frame: From day of first vaccination until 26 weeks after 3rd vaccination (study day 1 to day 211)
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 (PfSPZ Vaccine) | Arm 2 (Normal Saline)
Number analyzed (Participants) | 139 | 138
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Receipt of AL treatment to 26 weeks post 3rd vaccination (study day -17 to study day 211) = ~8 months
Arm/Group | Arm 1 (PfSPZ Vaccine) | Arm 2 (Normal Saline) | Enrolled With no Arm Assignment
All-Cause Mortality (participants affected / at risk) | 0/139 | 0/138 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/139 | 0/138 | 0/13
Other Adverse Events (participants affected / at risk) | 134/139 | 128/138 | 4/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (PfSPZ Vaccine) (N=139) | Arm 2 (Normal Saline) (N=138) | Enrolled With no Arm Assignment (N=13)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 10 (10) | 11 (12) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Bronchiolitis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 12 (12) | 10 (12) | 1 (1)
Conjunctivitis (Eye disorders) | 5 (5) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 20 (24) | 16 (18) | 0 (0)
Dental caries (Gastrointestinal disorders) | 2 (2) | 2 (3) | 0 (0)
Dermatosis (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
Ear infection (Infections and infestations) | 5 (5) | 4 (4) | 0 (0)
Eye injury (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0)
Face edema (General disorders) | 1 (1) | 0 (0) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 3 (3) | 6 (6) | 0 (0)
Forearm fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Furuncle (Infections and infestations) | 3 (3) | 4 (5) | 1 (1)
Gastroenteritis (Infections and infestations) | 5 (5) | 6 (6) | 0 (0)
Genitourinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 19 (21) | 22 (23) | 0 (0)
Hemoglobin decrease (Investigations) | 1 (1) | 0 (0) | 0 (0)
Hemoglobin increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Hernia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperleukocytosis (Blood and lymphatic system disorders) | 3 (3) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 6 (6) | 7 (8) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Malaria (Infections and infestations) | 86 (141) | 90 (146) | 0 (0)
Mumps (Infections and infestations) | 1 (1) | 3 (3) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 7 (7) | 2 (2) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 9 (11) | 22 (26) | 0 (0)
Otitis externa (Infections and infestations) | 1 (2) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Pruritus generalized (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pyoderma (Infections and infestations) | 2 (2) | 4 (4) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 62 (96) | 57 (83) | 0 (0)
Sinobronchitis (Infections and infestations) | 22 (29) | 23 (26) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (4) | 0 (0) | 0 (0)
Tinea infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Torticollis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Typhoid fever (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Varicella (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 20 (20) | 13 (14) | 0 (0)
Wound infection (Infections and infestations) | 7 (7) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-12-01): https://cdn.clinicaltrials.gov/large-docs/30/NCT04940130/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-18): https://cdn.clinicaltrials.gov/large-docs/30/NCT04940130/SAP_001.pdf